CLINICAL TRIAL: NCT04700449
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II Clinical Trial to Evaluate the Efficacy and Safety of CBP-307 in Subjects With Moderate to Severe Ulcerative Colitis (UC)
Brief Title: A Study Assessing the Efficacy and Safety of CBP-307 in Subjects With Moderate to Severe Ulcerative Colitis (UC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Connect Biopharm LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBP-307CN002
Record Dates: First submitted 2020-10-22; First posted 2021-01-07 (Actual); Results first posted 2023-11-02 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-04

CONDITIONS: Moderate to Severe Ulcerative Colitis
MeSH Terms: interventions — Double-Blind Method

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Double-Blind 0.2mg CBP-307 (Experimental): 0.2 mg CBP-307 capsules oral administration.
  Interventions: Drug: Double-Blind 0.2mg CBP-307
- Double-Blind Placebo (Placebo Comparator): Placebo capsules oral administration.
  Interventions: Drug: Double-Blind Placebo
- Open-Label CBP-307 (Experimental): 0.2 mg CBP-307 capsules oral administration.
  Interventions: Drug: Open-label CBP-307
- Double-Blind 0.1mg CBP-307 (Experimental): 0.1 mg CBP-307 capsules oral administration.
  Interventions: Drug: Double-Blind 0.1mg CBP-307

INTERVENTIONS:
Drug: Double-Blind 0.2mg CBP-307 — 0.2 mg capsule oral administration
  Arms: Double-Blind 0.2mg CBP-307
Drug: Double-Blind Placebo — Placebo capsule oral administration
  Arms: Double-Blind Placebo
Drug: Open-label CBP-307 — 0.2 mg capsule oral administration
  Arms: Open-Label CBP-307
Drug: Double-Blind 0.1mg CBP-307 — 0.1 mg capsule oral administration
  Arms: Double-Blind 0.1mg CBP-307

SUMMARY:
This study will evaluate the efficacy and safety of CBP-307 in subjects with moderate to severe ulcerative colitis (UC).

DETAILED DESCRIPTION:
This is a multicenter, multicountry, randomized, double-blind, placebo-controlled phase II clinical trial to evaluate the efficacy and safety of CBP-307 in subjects with moderate to severe ulcerative colitis (UC). CBP-307 capsules are administered orally. This study includes stage 1 and stage 2.

Study Stage 1 After screening, subjects entered the randomized, double-blind, placebo-controlled induction therapy for 12 weeks.

Subjects were screened at 1 to 21 days prior to the baseline visit. The eligible subjects were enrolled and randomized at the baseline visit. As per study protocol (version 5.0 or earlier), subjects received CBP 307 0.1 mg, CBP-307 0.2 mg, and placebo at a ratio of 1:1:1. The subjects enrolled under protocol (version 6.0) were randomized to CBP-307 0.2 mg and placebo at a ratio of 1:1 into the 2 groups (approximately 52 subjects in each group) and stratified according to whether the subject failed a previous tumor necrosis factor (TNF)-α antagonist therapy. Subjects assigned were blinded to their treatment assignment (CBP-307 or placebo) in the 12-week double-blinded placebo-controlled treatment period.

Subjects randomized to CBP-307 group underwent dose titration for 1 week, while those in placebo group underwent simulated titration. Both CBP-307 and placebo were administered through the oral route. For subjects in the CBP-307 0.1 mg QD group, a daily dose of 0.05 mg CBP-307 was given from Day 1 to Day 4; then a daily dose of 0.1 mg CBP-307 was given for 3 days from Day 5 to Day 7; from Day 8, a daily target dose of 0.1 mg was administered. For subjects in the group of CBP-307 0.2 mg QD, a daily dose of 0.05 mg CBP-307 was given from Day 1 to Day 4; then, a dose of 0.1 mg CBP-307 was given daily for 3 days from Day 5 to Day 7; from Day 8, a daily target dose of 0.2 mg was administered.

For the subjects already enrolled as per study protocol version 5.0 or earlier, they continued the treatment in the Stage 1 according to the previous planned schedule.

Eligible subjects completing 12 weeks of induction therapy in Stage 1 were permitted to enter Stage 2 to be evaluated for the long-term maintenance administration of CBP-307. Subjects who withdrew early from the study or completed the Stage 1, but did not enter Stage 2, entered a 4-week safety follow-up period.

Study stage 2 All subjects who completed 12 weeks of induction therapy in the study Stage 1 and completed all examinations (including colonoscopy) at Week 12 (visit 11) could choose to enter the study Stage 2 of a total length of 40 weeks, including 36 weeks of continuous treatment and 4 weeks of safety follow up after the last dose. Subjects who chose to enter the Stage 2 signed an updated informed consent form (ICF) and screened for eligibility.

The study Stage 2 contained sub-study 1 and sub-study 2. Subjects entered 1 of sub-studies based on their results of efficacy evaluation in the study Stage 1.

Sub-study 1 (subjects who achieved clinical response by adapted Mayo score): Subjects who achieved clinical response at Week 12 in the study Stage 1 and met the eligibility criteria for Stage 2 entered sub study 1 of the study Stage 2 to receive double-blind maintenance treatment for 36 weeks (Week 13 to 48), i.e., the therapeutic regimen for them in Stage 1 was continually maintained. Safety follow-up was completed at 4 weeks after the last dose. Subjects who presented with recurrent UC during maintenance treatment were terminated from the treatment and withdrew from the study.

For the subjects already enrolled as per study protocol version 5.0 or earlier, they followed the previous planned treatment in the sub-study 1 of Stage 2 study.

Sub-study 2 (subjects who did not achieve clinical response by adapted Mayo score): Subjects who did not achieve clinical response at Week 12 in study Stage 1 and met the eligibility criteria for Stage 2 entered open-label treatment with CBP-307 0.2 mg. Subjects received CBP-307 QD at an oral dose of 0.2 mg in sub study 2 regardless of whether they received CBP-307 or placebo in the study Stage 1.

For subjects who entered sub-study 2 of study Stage 2, 1-week dose titration was performed at Week 13. Dose titration involved administration of CBP 0.05 mg for 4 consecutive days from Titration Day 1 to Day 4, followed by administration of CBP-307 0.1 mg for 3 days from Titration Day 5 to Day 7, and administration of CBP-307 at a target dose of 0.2 mg initiated on Titration Day 8. After dose titration was completed, subjects received oral treatment with CBP-307 0.2 mg QD, for 36 weeks. Safety follow-up was completed at 4 weeks after the last dose. If the subjects did not achieve clinical response by the efficacy evaluation including colonoscopy at Week 24, the treatment was to be discontinued and the subjects were to withdraw from the study.

ELIGIBILITY:
Main inclusion and exclusion criteria for the study Stage 1:

Subjects were eligible to be included in the study only if all the following criteria applied:

* Male or female subjects aged 18 to 75 years (inclusive) with a diagnosis of UC established at least 3 months prior to screening by clinical and endoscopic evidence corroborated by a histopathology report;
* Confirmed to have moderately to severely active UC within 14 days prior to the first dose of the investigational product, based on an adapted Mayo score of 4 to 9, and an endoscopic subscore of ≥2;
* Had evidence of UC extending to the rectum with ≥15 cm involvement on endoscopy;
* UC patients who were receiving treatment. Subjects could be enrolled if they met any items below:

  1. Prior to the randomization visit, subjects had received oral 5-aminosalicylic acid (5-ASA) (e.g., mesalazine, sulfasalazine, olsalazine, balsalazide) for at least 4 weeks with the dose stable for at least 2 weeks;
  2. Prior to the randomization visit, subjects had received oral or intravenous (IV) corticosteroids e.g. prednisone (daily doses ≤30 mg), budesonide (daily doses ≤9 mg), methylprednisolone (daily doses ≤24 mg), or equivalent dose of corticosteroids for at least 4 weeks, with the dose stable for at least 2 weeks;
* Oral 5-ASA or corticosteroid for treatment of UC had been stopped for at least 2 weeks prior to the screening endoscopy examination which was used for Mayo score assessment;
* A stable dosing regimen had to be used if non-prohibited concomitant medications were used.

Subjects who met any of the following criteria were excluded:

* Subjects had evidence of toxic megacolon;
* Had subtotal or total colectomy;
* An existing ileostomy, colostomy, or known symptomatic stenosis of the intestine; a history or evidence of adenomatous colonic polyps that had not been removed; a history or evidence of colonic mucosal dysplasia including low or high grade of dysplasia, as well as indeterminate for dysplasia; a suspected or confirmed diagnosis of Crohn's enterocolitis, undiagnosed types of colitis, ischemic colitis, or radiation colitis;
* Previous exposure to lymphocyte-depleting therapies or D-penicillamine, leflunomide; prior exposure to approved or investigational products that inhibited the lymphocyte trafficking;
* Received immunosuppressants within 30 days prior to randomization; received any investigational biologic or non-biologic agent, or approved biologic agent or biosimilars within 60 days or 5 half lives prior to screening (whichever was longer);
* Known active infection during the screening period; treatment for Clostridioides difficile (C. difficile) infection or other intestinal pathogen with 28 days prior to first dose of investigational product; active or latent tuberculosis (TB); Chronic hepatitis B virus (HBV) infection or chronic hepatitis C virus (HCV) infection; any identified congenital or acquired immunodeficiency;
* Received any live vaccine within 30 days prior to screening.

Main Inclusion and exclusion criteria for subjects' entry into the study Stage 2 from Stage 1:

Subjects who met all the following criteria entered into the study Stage 2:

* subjects with UC who completed 12 weeks of treatment with CBP-307 or placebo in Stage 1 and completed all the assessments (including colonoscopy) at study visit of Week 12 in study Stage 1;
* Good compliance in Stage 1;
* Subjects or their legal representatives voluntarily signed the ICF for study Stage 2.

Subjects who met any of the following criteria were excluded from the study Stage 2:

* subjects had any unstable or uncontrolled cardiovascular, pulmonary, hepatic, renal, gastrointestinal, genitourinary, hematological, coagulation, immunological, endocrine/metabolic, or other medical disorder that, in the opinion of the investigator, were to confound the study results or compromise subject safety;
* Allergic to CBP 307 or its excipients, experience of significant adverse events related to the study drug during Stage 1, and not appropriate to participate in Stage 2 assessed by the investigator;
* Active or chronic recurrent infections;
* A history of uveitis or macular oedema.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2022-02-23 (Actual); Study Completion 2022-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzhou Connect, Study Director — Connect Biopharm LLC
Locations (66):
- United States (14):
  - Connect Investigative Site 2316, Phoenix, Arizona
  - Connect Investigative Site 2308, Mission Hills, California
  - Connect Investigative Site 2314, Hialeah, Florida
  - Connect Investigative Site 2309, Homestead, Florida
  - Connect Investigative Site 2320, Kissimmee, Florida
  - Connect Investigative Site 2318, Miami, Florida
  - Connect Investigative Site 2302, Orlando, Florida
  - Connect Investigative Site 2304, Orlando, Florida
  - Connect Investigative Site 2306, Orlando, Florida
  - Connect Investigative Site 2307, Atlanta, Georgia
  - Connect Investigative Site 2315, Cincinnati, Ohio
  - Connect Investigative Site 2321, Oklahoma City, Oklahoma
  - Connect Investigative Site 2311, Cypress, Texas
  - Connect Investigative Site 2319, San Antonio, Texas
- China (39):
  - Connect Investigative Site 2018, Hefei, Anhui
  - Connect Investigative Site 2004, Hefei, Anhui
  - Connect Investigative Site 2008, Beijing, Beijing Municipality
  - Connect Investigative Site 2001, Beijing, Beijing Municipality
  - Connect Investigative Site 2015, Jilin, Changchun
  - Connect Investigative Site 2006, Fuzhou, Fujian
  - Connect Investigative Site 2012, Xiamen, Fujian
  - Connect Investigative Site 2003, Guangzhou, Guangdong
  - Connect Investigative Site 2009, Guangzhou, Guangdong
  - Connect Investigative Site 2017, Shenzhen, Guangdong
  - Connect Investigative Site 2021, Shenzhen, Guangdong
  - Connect Investigative Site 2030, Nanning, Guangxi
  - Connect Investigative Site 2034, Haikou, Hainan
  - Connect Investigative Site 2026, Shijiazhuang, Hebei
  - Connect Investigative Site 2041, Shijiazhuang, Hebei
  - Connect Investigative Site 2022, Zhengzhou, Henan
  - Connect Investigative Site 2016, Wuhan, Hubei
  - Connect Investigative Site 2005, Wuhan, Hubei
  - Connect Investigative Site 2027, Nanjing, Jiangsu
  - Connect Investigative Site 2031, Nanjing, Jiangsu
  - Connect Investigative Site 2023, Nanjing, Jiangsu
  - Connect Investigative Site 2033, Suzhou, Jiangsu
  - Connect Investigative Site 2046, Nanchang, Jiangxi
  - Connect Investigative Site 2025, Dalian, Liaoning
  - Connect Investigative Site 2040, Shenyang, Liaoning
  - Connect Investigative Site 2028, Jinan, Shandong
  - Connect Investigative Site 2044, Jinan, Shandong
  - Connect Investigative Site 2024, Qingdao, Shandong
  - Connect Investigative Site 2011, Shanghai, Shanghai Municipality
  - Connect Investigative Site 2007, Shanghai, Shanghai Municipality
  - Connect Investigative Site 2019, Shanghai, Shanghai Municipality
  - Connect Investigative Site 2035, Shanghai, Shanghai Municipality
  - Connect Investigative Site 2038, Shanghai, Shanghai Municipality
  - Connect Investigative Site 2020, Taiyuan, Shanxi
  - Connect Investigative Site 2013, Chengdu, Sichuan
  - Connect Investigative Site 2043, Chongqing, Sichuan
  - Connect Investigative Site 2047, Hangzhou, Zhejiang
  - Connect Investigative Site 2032, Hangzhou, Zhejiang
  - Connect Investigative Site 2045, Wenzhou, Zhejiang
- Pakistan (2):
  - Connect Investigative Site 2151, Karachi, Sindh
  - Connect Investigative Site 2152, Karachi, Sindh
- Ukraine (11):
  - Connect Investigative Site 2211, Dnipro
  - Connect Investigative Site 2217, Ivano-Frankivsk
  - Connect Investigative Site 2202, Kharkiv
  - Connect Investigative Site 2208, Kharkiv
  - Connect Investigative Site 2205, Kyiv
  - Connect Investigative Site 2220, Kyiv
  - Connect Investigative Site 2215, Lviv
  - Connect Investigative Site 2216, Lviv
  - Connect Investigative Site 2218, Uzhhorod
  - Connect Investigative Site 2209, Vinnytsia
  - Connect Investigative Site 2214, Zaporizhzhia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Because 1 subject in stage 1 placebo group was randomized but not treated, so the Enrollment number in the Protocol Section (145) conflicts with the number of participants Started in the Participant Flow module (144).
Groups:
- Double-Blind 0.1 mg CBP-307: 0.1 mg CBP-307 capsules oral administration.
- Double-Blind 0.2 mg CBP-307: 0.2 mg CBP-307 capsules oral administration.
- Double-Blind Placebo: Placebo capsules oral administration.
  Placebo: Placebo capsules oral administration
- Open-Label 0.2 mg CBP-307: 0.2 mg CBP-307 capsule oral administration
Period: Stage 1: Double-Blind Period
Arm/Group | Double-Blind 0.1 mg CBP-307 | Double-Blind 0.2 mg CBP-307 | Double-Blind Placebo | Open-Label 0.2 mg CBP-307
Started | 39 | 53 | 52 | 0
Completed | 28 | 50 | 47 | 0
Not Completed | 11 | 3 | 5 | 0
Not completed — Adverse Event | 5 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 2 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0
Not completed — COVID-19 Restriction | 3 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 1 | 0
Period: Stage 2 Sub-study 1
Arm/Group | Double-Blind 0.1 mg CBP-307 | Double-Blind 0.2 mg CBP-307 | Double-Blind Placebo | Open-Label 0.2 mg CBP-307
Started | 12 | 21 | 13 | 0
Completed | 10 | 17 | 9 | 0
Not Completed | 2 | 4 | 4 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 2 | 0
Not completed — COVID-19 Restriction | 0 | 0 | 1 | 0
Not completed — Other | 1 | 2 | 0 | 0
Period: Stage 2 Sub-study 2
Arm/Group | Double-Blind 0.1 mg CBP-307 | Double-Blind 0.2 mg CBP-307 | Double-Blind Placebo | Open-Label 0.2 mg CBP-307
Started | 0 | 0 | 0 | 40
Completed | 0 | 0 | 0 | 17
Not Completed | 0 | 0 | 0 | 23
Not completed — Adverse Event | 0 | 0 | 0 | 7
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 9
Not completed — COVID-19 Restriction | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 5

BASELINE CHARACTERISTICS:
Population: Because 1 subject in stage 1 placebo group was randomized but not treated, so the Overall Number of Baseline Participants in "Double-Blind Placebo" is greater than the number of participants included in the Participant Flow module.
Groups:
- Total: Total of all reporting groups
Arm/Group | Double-Blind 0.1 mg CBP-307 | Double-Blind 0.2 mg CBP-307 | Double-Blind Placebo | Total
Number analyzed (Participants) | 39 | 53 | 53 | 145
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Demographic and Other Baseline Characteristics (Stage 1) - Randomized Set
  years | 42.9 (13.41) | 42.1 (10.66) | 41.2 (9.86) | 42 (11.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 20 | 20 | 54
  Male | 25 | 33 | 33 | 91
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 39 | 48 | 46 | 133
  Black or African American | 0 | 0 | 1 | 1
  White | 0 | 5 | 4 | 9
  Not Reported | 0 | 0 | 2 | 2
  Hispanic or Latino | 0 | 1 | 3 | 4
  Not Hispanic or Latino | 39 | 52 | 50 | 141
Adapt Mayo Score at Baseline [Mean (Standard Deviation); unit: units on a scale] — Adapted Mayo scores were calculated based on data in stool frequency, rectal bleeding, and endoscopic findings. The Mayo scores range from 0 to 9 and consist of 3 subscores, each ranging from 0 to 3. The higher the score is, the more severe the disease is.
  units on a scale | 6.00 (1.485) | 5.84 (1.361) | 5.93 (1.178) | 5.92 (1.325)
Complete Mayo Score at Baseline [Mean (Standard Deviation); unit: units on a scale] — Complete Mayo scores were calculated based on data in stool frequency, rectal bleeding, endoscopic findings, and physician's global assessment. The Mayo scores range from 0 to 12 and consist of 4 subscores, each ranging from 0 to 3. The higher the score is, the more severe the disease is.
  units on a scale | 8.15 (1.641) | 8.03 (1.518) | 8.12 (1.282) | 8.10 (1.463)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline for Adapted Mayo Score: 0.2 mg Versus Placebo
Description: Change in adapted Mayo score from baseline at week 12 compared between CBP-307 0.2 mg and placebo in the Full Analysis Set by Multiple Imputation. Adapted Mayo scores were calculated based on data in stool frequency, rectal bleeding, and endoscopic findings. The Mayo scores range from 0 to 9 and consist of 3 subscores, each ranging from 0 to 3. The higher the score is, the more severe the disease is.
Time Frame: The adapted Mayo score was evaluated at screening and Week 12 (or early termination visit) during the study Stage 1 as well as at Week 24 (only for the sub-study 2) and Week 48 (or early termination visit) during the study Stage 2.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Double-Blind 0.2 mg CBP-307 | Double-Blind Placebo
Number analyzed (Participants) | 53 | 52
score on a scale | -2.60 [-3.716 to -1.477] | -1.95 [-3.073 to -0.834]

2. Secondary Outcome: Change in Complete Mayo Score From Baseline
Description: Change in complete Mayo score from baseline at week 12 after treatment. Complete Mayo scores were calculated based on data in stool frequency, rectal bleeding, endoscopic findings, and physician's global assessment. The Mayo scores range from 0 to 12 and consist of 4 subscores, each ranging from 0 to 3. The higher the score is, the more severe the disease is.
Time Frame: at Week 12
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Double-Blind 0.1 mg CBP-307 | Double-Blind 0.2 mg CBP-307 | Double-Blind Placebo
Number analyzed (Participants) | 39 | 53 | 52
score on a scale | -3.87 [-5.407 to -2.324] | -3.67 [-4.959 to -2.385] | -2.74 [-4.030 to -1.458]

3. Secondary Outcome: Comparison of Clinical Response Rate by Adapted Mayo Score
Description: Comparison of clinical response rate at week 12 by adapted Mayo score (defined as a decrease of ≥ 2 points and at least 30% from baseline, accompanied with a decrease of ≥ 1 point from baseline in the rectal bleeding subscore or an absolute rectal bleeding subscore of ≤ 1 point).
Time Frame: at Week 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Double-Blind 0.1 mg CBP-307 | Double-Blind 0.2 mg CBP-307 | Double-Blind Placebo
Number analyzed (Participants) | 39 | 53 | 52
percentage of participants | 35.9 [20.84 to 50.95] | 52.8 [39.39 to 66.27] | 32.7 [19.94 to 45.44]

4. Secondary Outcome: Comparison of Clinical Response Rate by Complete Mayo Score
Description: Comparison of clinical response rate at week 12 by complete Mayo score (defined as a decrease of ≥ 3 points and at least 30% from baseline, accompanied with a decrease of ≥ 1 point from baseline in the rectal bleeding subscore or an absolute rectal bleeding subscore of ≤ 1 point).
Time Frame: at Week 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Double-Blind 0.1 mg CBP-307 | Double-Blind 0.2 mg CBP-307 | Double-Blind Placebo
Number analyzed (Participants) | 39 | 53 | 52
percentage of participants | 35.9 [20.84 to 50.95] | 50.9 [37.48 to 64.40] | 28.8 [16.53 to 41.16]

5. Secondary Outcome: Comparison of Clinical Remission Rate by Adapted Mayo Score
Description: Comparison of clinical remission rate at week 12 by adapted Mayo score (defined as a rectal bleeding subscore = 0 and a stool frequency subscore ≤ 1, with an Endoscopy subscore ≤ 1 [excluding friability]).
Time Frame: at Week 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Double-Blind 0.1 mg CBP-307 | Double-Blind 0.2 mg CBP-307 | Double-Blind Placebo
Number analyzed (Participants) | 39 | 53 | 52
percentage of participants | 12.8 [2.33 to 23.31] | 28.3 [16.17 to 40.43] | 9.6 [1.60 to 17.63]

6. Secondary Outcome: Comparison of Clinical Remission Rate by Complete Mayo Score
Description: Comparison of clinical remission rate at week 12 by complete Mayo score (defined as a total Mayo score of ≤ 2 points with no individual subscore > 1 point).
Time Frame: at Week 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Double-Blind 0.1 mg CBP-307 | Double-Blind 0.2 mg CBP-307 | Double-Blind Placebo
Number analyzed (Participants) | 39 | 53 | 52
percentage of participants | 10.3 [0.73 to 19.78] | 20.8 [9.84 to 31.67] | 5.8 [0.00 to 12.11]

7. Secondary Outcome: Mucosal Healing Rate
Description: Mucosal healing rate at week 12 after treatment (mucosal healing is defined as Mayo endoscopic subscore ≤ 1)
Time Frame: at Week 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Double-Blind 0.1 mg CBP-307 | Double-Blind 0.2 mg CBP-307 | Double-Blind Placebo
Number analyzed (Participants) | 39 | 53 | 52
percentage of participants | 20.5 [7.84 to 33.19] | 30.2 [17.83 to 42.55] | 21.2 [10.05 to 32.25]

8. Secondary Outcome: Incidence, Type and Severity of Treatment Emergent Adverse Event (TEAE)
Description: The safety and tolerability will be assessed on basis of incidence, type and severity of TEAEs as well as their relations with the investigational product .
Time Frame: for 12 consecutive weeks
Measure: Number; unit: cases
Groups:
- Stage 1 Double-Blind 0.1 mg CBP-307; Stage 2 Double-Blind 0.1 mg CBP-307: 0.1 mg CBP-307 capsules oral administration.
- Stage 1 Double-Blind 0.2 mg CBP-307; Stage 2 Double-Blind 0.2 mg CBP-307; Stage 2 Open-label 0.2 mg CBP-307: 0.2 mg CBP-307 capsules oral administration.
- Stage 1 Double-Blind Placebo; Stage 2 Double-Blind Placebo: Placebo capsules oral administration.
Arm/Group | Stage 1 Double-Blind 0.1 mg CBP-307 | Stage 1 Double-Blind 0.2 mg CBP-307 | Stage 1 Double-Blind Placebo | Stage 2 Double-Blind 0.1 mg CBP-307 | Stage 2 Double-Blind 0.2 mg CBP-307 | Stage 2 Double-Blind Placebo | Stage 2 Open-label 0.2 mg CBP-307
Number analyzed (Participants) | 39 | 53 | 52 | 12 | 21 | 13 | 40
cases
  Gastrointestinal disorders | 12 | 16 | 14 | 4 | 11 | 3 | 17
  Infections and infestations | 14 | 13 | 15 | 2 | 6 | 6 | 10
  Investigations | 13 | 18 | 9 | 5 | 9 | 3 | 13
  Cardiac disorders | 9 | 13 | 6 | 4 | 4 | 2 | 6
  Eye disorders | 5 | 11 | 10 | 5 | 7 | 5 | 5
  Nervous system disorders | 6 | 8 | 9 | 1 | 5 | 1 | 2
  Skin and subcutaneous tissue disorders | 9 | 5 | 4 | 5 | 2 | 1 | 3
  Blood and lymphatic system disorders | 6 | 4 | 8 | 1 | 3 | 0 | 5
  Respiratory, thoracic and mediastinal disorders | 6 | 6 | 5 | 3 | 5 | 1 | 4
  General disorders and administration site conditions | 5 | 7 | 4 | 1 | 4 | 0 | 5
  Metabolism and nutrition disorders | 4 | 7 | 3 | 2 | 4 | 1 | 3
  Hepatobiliary disorders | 7 | 5 | 1 | 3 | 3 | 1 | 4
  Musculoskeletal and connective tissue disorders | 2 | 5 | 2 | 2 | 5 | 2 | 3
  Vascular disorders | 0 | 3 | 3 | 1 | 2 | 0 | 0
  Renal and urinary disorders | 3 | 1 | 1 | 0 | 0 | 1 | 2
  Injury, poisoning and procedural complications | 2 | 1 | 0 | 1 | 1 | 0 | 0
  Psychiatric disorders | 1 | 2 | 0 | 0 | 2 | 0 | 2
  Reproductive system and breast disorders | 0 | 1 | 1 | 0 | 1 | 1 | 0
  Ear and labyrinth disorders | 1 | 1 | 1 | 1 | 0 | 0 | 1

9. Secondary Outcome: Incidence, Type and Severity of Serious Adverse Event (SAE)
Description: The safety and tolerability will be assessed on basis of incidence, type and severity of SAEs as well as their relations with the investigational product and SAEs that lead to discontinuation of study.
Time Frame: for 12 consecutive weeks
Measure: Number; unit: cases
Arm/Group | Stage 1 Double-Blind 0.1 mg CBP-307 | Stage 1 Double-Blind 0.2 mg CBP-307 | Stage 1 Double-Blind Placebo | Stage 2 Double-Blind 0.1 mg CBP-307 | Stage 2 Double-Blind 0.2 mg CBP-307 | Stage 2 Double-Blind Placebo | Stage 2 Open-label 0.2 mg CBP-307
Number analyzed (Participants) | 39 | 53 | 52 | 12 | 21 | 13 | 40
cases
  Colitis ulcerative | 4 | 2 | 2 | 0 | 0 | 0 | 6
  Gastritis | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Transitional cell carcinoma | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Ovarian cyst | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Appendicitis | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Large intestine polyp | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Anal abscess | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Cholera | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Cytomegalovirus infection | 0 | 0 | 0 | 0 | 0 | 0 | 1

10. Secondary Outcome: Incidence, Type and Severity of Adverse Events (AE)
Description: The safety and tolerability will be assessed on basis of AEs that lead to discontinuation of study, and AEs of special interest (cardiac events as well as pulmonary function tests, ophthalmologic examinations, skin examinations, and nervous system physical examinations)
Time Frame: for 12 consecutive weeks
Population: Treatment-Emergent Adverse Events Leading to Study Drug Withdrawal
Measure: Number; unit: cases
Arm/Group | Stage 1 Double-Blind 0.1 mg CBP-307 | Stage 1 Double-Blind 0.2 mg CBP-307 | Stage 1 Double-Blind Placebo | Stage 2 Double-Blind 0.1 mg CBP-307 | Stage 2 Double-Blind 0.2 mg CBP-307 | Stage 2 Double-Blind Placebo | Stage 2 Open-label 0.2 mg CBP-307
Number analyzed (Participants) | 39 | 53 | 52 | 12 | 21 | 13 | 40
cases
  Hepatobiliary disorders (Leading to Drug Withdrawal) | 4 | 0 | 0 | 0 | 0 | 0 | 0
  Eye disorders (Leading to Drug Withdrawal) | 1 | 1 | 0 | 0 | 1 | 0 | 1
  Gastrointestinal disorders (Leading to Drug Withdrawal) | 0 | 1 | 0 | 0 | 0 | 0 | 3
  Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Leading to Drug Withdrawal) | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Infections and infestations (Leading to Drug Withdrawal) | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Hepatobiliary disorders (Treatment-Emergent Adverse Events of Special Interest) | 4 | 0 | 0 | 0 | 0 | 0 | 1
  Cardiac disorders (Treatment-Emergent Adverse Events of Special Interest) | 1 | 1 | 0 | 0 | 1 | 0 | 2
  Eye disorders (Treatment-Emergent Adverse Events of Special Interest) | 1 | 1 | 0 | 0 | 1 | 0 | 1
  Respiratory disorders (Treatment-Emergent Adverse Events of Special Interest) | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Investigations (Treatment-Emergent Adverse Events of Special Interest) | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Infections and infestations (Treatment-Emergent Adverse Events of Special Interest) | 0 | 0 | 0 | 0 | 0 | 1 | 1

11. Secondary Outcome: Change From Baseline in Adapted Mayo Score: 0.1 mg Versus Placebo
Description: Change from baseline in adapted Mayo score at Week 12 between CBP-307 0.1 mg and placebo in the Full Analysis Set by Multiple Imputation. Adapted Mayo scores were calculated based on data in stool frequency, rectal bleeding, and endoscopic findings. The Mayo scores range from 0 to 9 and consist of 3 subscores, each ranging from 0 to 3. The higher the score is, the more severe the disease is.
Time Frame: at Week 12
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Double-Blind Placebo: Placebo: Placebo capsules oral administration
Arm/Group | Double-Blind 0.1 mg CBP-307 | Double-Blind Placebo
Number analyzed (Participants) | 39 | 52
score on a scale | -2.90 [-4.121 to -1.679] | -1.95 [-3.073 to -0.834]

ADVERSE EVENTS:
Time Frame: Adverse events were persistently monitored throughout the study, from the time of informed consent until 28 days after the last dose, up to 55 weeks.
Arm/Group | Stage 1 Double-Blind 0.1 mg CBP-307 | Stage 1 Double-Blind 0.2 mg CBP-307 | Stage 1 Double-Blind Placebo | Stage 2 Double-Blind 0.1 mg CBP-307 | Stage 2 Double-Blind 0.2 mg CBP-307 | Stage 2 Double-Blind Placebo | Stage 2 Open-label 0.2 mg CBP-307
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/53 | 0/52 | 0/12 | 0/21 | 0/13 | 0/40
Serious Adverse Events (participants affected / at risk) | 6/39 | 2/53 | 3/52 | 0/12 | 1/21 | 0/13 | 8/40
Other Adverse Events (participants affected / at risk) | 37/39 | 47/53 | 40/52 | 11/12 | 20/21 | 12/13 | 33/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1 Double-Blind 0.1 mg CBP-307 (N=39) | Stage 1 Double-Blind 0.2 mg CBP-307 (N=53) | Stage 1 Double-Blind Placebo (N=52) | Stage 2 Double-Blind 0.1 mg CBP-307 (N=12) | Stage 2 Double-Blind 0.2 mg CBP-307 (N=21) | Stage 2 Double-Blind Placebo (N=13) | Stage 2 Open-label 0.2 mg CBP-307 (N=40)
Colitis ulcerative (Gastrointestinal disorders) | 4 | 2 | 2 | 0 | 0 | 0 | 6
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholera (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1 Double-Blind 0.1 mg CBP-307 (N=39) | Stage 1 Double-Blind 0.2 mg CBP-307 (N=53) | Stage 1 Double-Blind Placebo (N=52) | Stage 2 Double-Blind 0.1 mg CBP-307 (N=12) | Stage 2 Double-Blind 0.2 mg CBP-307 (N=21) | Stage 2 Double-Blind Placebo (N=13) | Stage 2 Open-label 0.2 mg CBP-307 (N=40)
Gastrointestinal disorders (Gastrointestinal disorders) | 12 | 16 | 14 | 4 | 11 | 3 | 17
Infections and infestations (Infections and infestations) | 14 | 13 | 15 | 2 | 6 | 6 | 10
Investigations (Investigations) | 13 | 18 | 9 | 5 | 9 | 3 | 13
Cardiac disorders (Cardiac disorders) | 9 | 13 | 6 | 4 | 4 | 2 | 6
Eye disorders (Eye disorders) | 5 | 11 | 10 | 5 | 7 | 5 | 5
Nervous system disorders (Nervous system disorders) | 6 | 8 | 9 | 1 | 5 | 1 | 2
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 9 | 5 | 4 | 5 | 2 | 1 | 3
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 6 | 4 | 8 | 1 | 3 | 0 | 5
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 6 | 6 | 5 | 3 | 5 | 1 | 4
General disorders and administration site conditions (General disorders) | 5 | 7 | 4 | 1 | 4 | 0 | 5
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 4 | 7 | 3 | 2 | 4 | 1 | 3
Hepatobiliary disorders (Hepatobiliary disorders) | 7 | 5 | 1 | 3 | 3 | 1 | 4
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 2 | 5 | 2 | 2 | 5 | 2 | 3
Vascular disorders (Vascular disorders) | 0 | 3 | 3 | 1 | 2 | 0 | 0
Renal and urinary disorders (Renal and urinary disorders) | 3 | 1 | 1 | 0 | 0 | 1 | 2
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 1 | 1 | 0 | 0
Psychiatric disorders (Psychiatric disorders) | 1 | 2 | 0 | 0 | 2 | 0 | 2
Reproductive system and breast disorders (Reproductive system and breast disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 0
Ear and labyrinth disorders (Ear and labyrinth disorders) | 1 | 1 | 1 | 1 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-12-25): https://cdn.clinicaltrials.gov/large-docs/49/NCT04700449/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-18): https://cdn.clinicaltrials.gov/large-docs/49/NCT04700449/SAP_001.pdf